CLINICAL TRIAL: NCT00172744
Title: Effect of Cyclic Tensional Force on Osteogenic Differentiation of Human Periodontal Ligament Stem Cells
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701291
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2007-10-11 (Estimated); Status verified 2005-03

CONDITIONS: Healthy
Keywords: stem cells; periodontal cells; mechanical stress; differentiation; periodontal ligament

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to observe cyclic tensional force on the osteogenic differentiation of human periodontal ligament stem cells.

DETAILED DESCRIPTION:
This study is to investigate the effect of the cyclic mechanical strain on the osteogenic differentiation of mesenchymal stem cells. Mesenchymal stem cells will be cultured from the periodontal ligament tissue of the premolars extracted due to orthodontic reason.

ELIGIBILITY:
Inclusion Criteria:

* Orthodontic patients who need to have premolars extracted

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-04; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Jane Chen, MSD, Principal Investigator — School of Dentistry, College of Medicine, National Taiwan University
Locations (1):
- School of Dentistry, College of Medicine, National Taiwan University, Taipei, Taiwan